CLINICAL TRIAL: NCT01791803
Title: Smoking Cessation Treatment of CardioPulmonary Hospitalized Patients
Brief Title: Smoking Cessation After Hospitalization for a Cardiopulmonary Illness
Acronym: STOPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Shore Medical Center (Other)
Responsible Party: Principal Investigator, Faysal M. Hasan, MD, Director, Tobacco Prevention Service, North Shore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STOPP
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Tobacco abstinence; hypnotherapy; Nicotine replacement therapy
MeSH Terms: conditions — Smoking Cessation | interventions — Hypnosis; Nicotine; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Hypnotherapy (Experimental): Patients admitted with a cardiopulmonary illness received a 90 minute free hypnotherapy session within 2 weeks of discharge, and a standardized tape for smoking cessation and relaxation for continued use after the session. They also received self-help brochures, and counseling during hospitalization and by telephone at 1,2,4,8 and 12 weeks after discharge.
  Interventions: Behavioral: hypnotherapy
- Nicotine Replacement Therapy (Experimental): Patients recieved a free one month supply of Nicotine replacement therapy to include patches and Gum, lozenges or sprays. Patients also received self-help brochures, and counseling during hospitalization and by telephone at 1,2,4,8 and 12 weeks after hospitalization.
  Interventions: Drug: Nicotine
- Hypnotherapy and Nicotine replacement (Experimental): The group received similar hypnotherapy session and tape, similar brochure and counseling protocol, as well as free nicotine replacement supplies for a month after discharge.
  Interventions: Behavioral: hypnotherapy; Drug: Nicotine
- Self-Quit group (No Intervention): Patients were given brief counseling during hospitalization and will not be contacted until 26 weeks after hospitalization.

INTERVENTIONS:
Behavioral: hypnotherapy — One 90 minute session within 2 weeks of hospital discharge
  Other Names: hypnosis
  Arms: Hypnotherapy; Hypnotherapy and Nicotine replacement
Drug: Nicotine — free one month supply after hospital discharge
  Other Names: Nicotine replacement therapy
  Arms: Hypnotherapy and Nicotine replacement; Nicotine Replacement Therapy

SUMMARY:
Smoking-related cardiopulmonary diseases account for a large number of hospital admissions. We investigated the efficacy of hypnotherapy as an aid to a counseling-based smoking cessation program in improving quit rates of hospitalized smoking patients at 12 and 26 weeks after hospital discharge. We compared outcomes with hospitalized patients who received more conventional therapy, namely nicotine replacement therapy, or patients who decided to quit on their own. We also compared smoking cessation rates at 12 and 26 weeks after hospitalization among patients admitted with a cardiac or a pulmonary diagnosis.

DETAILED DESCRIPTION:
Hospitalized patients with a cardiopulmonary diagnosis who were contemplating quitting were recruited into 4 groups: Hypnotherapy, Nicotine replacement therapy (NRT), both hypnotherapy and NRT, and self-quit group. All patients received self-help brochures and in-hospital counseling. Intervention groups received more extensive counseling, free NRT supply for a month and/or a 90 minute hypnotherapy session within 2 weeks of discharge. They also had follow up telephone counseling at 1,2,4,8 and 12 weeks after discharge. 7 day prevalence of tobacco abstinence rates at 26 weeks after hospitalization were verified by self report and urinary Cotinine levels.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with a Cardiopulmonary admission.

Exclusion Criteria:

* Terminal illness, history of Serious Psychiatric illness or substance abuse, Pregnancy, Cognitive or language barriers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2006-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faysal Hasan, M.D., Principal Investigator — North Shore Medical Center
Locations (1):
- North Shore Medical Center, Salem, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
published in: Complementary Therapies in Medicine 2014: 22: 1-8.

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypnotherapy: Patients admitted with a cardiopulmonary illness will receive a 90 minute free hypnotherapy session within 2 weeks of discharge, and a standardized tape for smoking cessation and relaxation for continued use after the session. They will also recieve self-help brochures, and counseling during hospitalization and by telephone at 1,2,4,8 and 12 weeks after discharge.
  hypnotherapy: One 90 minute session within 2 weeks of hospital discharge
- Nicotine Replacement Therapy: Patients will recieve a free one month supply of Nicotine replacement therapy to include patches and Gum, lozenges or sprays. Patients will receive self-help brochures, and counseling during hospitalization and by telephone at 1,2,4,8 and 12 weeks after hospitalization.
  Nicotine: free one month supply after hospital discharge
- Hypnotherapy and Nicotine Replacement: The group will recieve similar hypnotherapy session and tape, similar brochure and counseling protocol, as well as free nictotine replacement supplies for a month after discharge.
  hypnotherapy: One 90 minute session within 2 weeks of hospital discharge
  Nicotine: free one month supply after hospital discharge
- Self-Quit Group: patients will be given brief counseling during hospitalization and will not be contacted until 26 weeks after hospitalization.
Period: Overall Study
Arm/Group | Hypnotherapy | Nicotine Replacement Therapy | Hypnotherapy and Nicotine Replacement | Self-Quit Group
Started | 41 | 41 | 40 | 42
Completed | 41 | 39 | 38 | 37
Not Completed | 0 | 2 | 2 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 2 | 0 | 1
Not completed — Death | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: patients included in analysis were less than numbers recruited in groups because some patients were eliminated due to severity of illness including mortality and one developed psychosis, thus became eligible. All patients that were lost to follow up were considered to be smokers for analysis.
Groups:
- Hypnotherapy: Patients received a 90 minute free hypnotherapy session within 2 weeks of discharge, and a standardized tape for smoking cessation and relaxation for continued use . They also received counseling during hospitalization and by telephone at 1,2,4,8 and 12 weeks after discharge.
- Nicotine Replacement Therapy: Patients received a free one month supply of Nicotine replacement therapy to include patches and Gum, lozenges or sprays, self-help brochures, and counseling during hospitalization and by telephone at 1,2,4,8 and 12 weeks after hospitalization.
- Hypnotherapy and Nicotine Replacement: patients recieved both a similar hypnotherapy session and tape, similar brochure and counseling protocol, as well as free nictotine replacement supplies for a month after discharge.
- Self-Quit Group: Patients were given brief counseling during hospitalization and were not contacted until 26 weeks after hospitalization. They received no telephone contact and or counseling after discharge.
- Total: Total of all reporting groups
Arm/Group | Hypnotherapy | Nicotine Replacement Therapy | Hypnotherapy and Nicotine Replacement | Self-Quit Group | Total
Number analyzed (Participants) | 41 | 41 | 40 | 42 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 41 | 41 | 40 | 42 | 164
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (10.6) | 55.3 (12.2) | 54.4 (8.9) | 56.0 (10.7) | 55.17 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 14 | 16 | 73
  Male | 16 | 23 | 26 | 26 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants] — White Race ( n, %)
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0
    White | 38 | 32 | 31 | 36 | 137
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 3 | 9 | 9 | 6 | 27
Region of Enrollment [Number; unit: participants]
  United States | 41 | 41 | 40 | 42 | 164
Years of education [Mean (Standard Deviation); unit: years] | 13 (2) | 12.6 (2) | 13.2 (1.8) | 13.2 (1.9) | 13 (1.9)
Number of cigarettes smoked [Mean (Standard Deviation); unit: Cigarettes smoked /day] | 19.8 (12.6) | 21.2 (12.6) | 20.5 (9.3) | 15 (10) | 19.12 (11.12)
Total years of smoking [Mean (Standard Deviation); unit: years] | 36.5 (12.7) | 34.2 (14.4) | 34.3 (11.7) | 33.2 (10.8) | 34.55 (12.4)
Living with a smoker [Count of Participants; unit: Participants] | 18 | 16 | 13 | 14 | 61
Admitted with Cardiac Diagnosis [Count of Participants; unit: Participants] | 26 | 25 | 22 | 27 | 100
Lost to Follow up (Considered non-quitters) [Count of Participants; unit: Participants] | 14 | 12 | 13 | 17 | 56

OUTCOME MEASURES:

1. Primary Outcome: Abstinence From Smoking
Description: Assessed by 7-day prevalence of verified tobacco abstinence at 26 weeks after hospitalization for a cardiopulmoanry illness. Verification was confirmed biochemically by urine Cotinine testing or by telephone and discussion with a household proxy. Patients lost to follow up were considered to be persistent smokers.
Time Frame: at 26 weeks after hospitalization
Measure: Number; unit: percentage of participants
Groups:
- Nicotine Replacement Therapy: Patients received a free one month supply of Nicotine replacement therapy to include patches and Gum, lozenges or sprays. Patients also received self-help brochures, and counseling during hospitalization and by telephone at 1,2,4,8 and 12 weeks after hospitalization.
  Nicotine: free one month supply after hospital discharge
Arm/Group | Hypnotherapy | Nicotine Replacement Therapy | Hypnotherapy and Nicotine Replacement | Self-Quit Group
Number analyzed (Participants) | 41 | 39 | 38 | 37
percentage of participants | 15 | 7 | 13 | 10
Statistical Analysis 1: Comparison: Hypnotherapy vs Nicotine Replacement Therapy; Test type: Superiority or Other; Risk Ratio (RR) = 2.6, 95% CI 2-sided [1.1 to 11.4]
Statistical Analysis 2: Comparison: Nicotine Replacement Therapy vs Hypnotherapy and Nicotine Replacement; Test type: Superiority or Other; Risk Ratio (RR) = 2.4, 95% CI 2-sided [1.04 to 9.7]

2. Secondary Outcome: Smoking Cessation
Description: Abstinence from smoking at 12 weeks after hospitalization was measured by self reported 7-day prevalence and verified urinary Cotinine test. This included participants in groups receiving hypnotherapy, NRT or both. Self quit group was not approached until 26 weeks after discharge. Patients lost to follow up were considered smokers.
Time Frame: at 12 weeks after hospitalization
Measure: Count of Participants; unit: Participants
Groups:
- Hypnotherapy: Patients admitted with a cardiopulmonary illness received a 90 minute free hypnotherapy session within 2 weeks of discharge, and a standardized tape for smoking cessation and relaxation for continued use after the session. They will also recieve self-help brochures, and counseling during hospitalization and by telephone at 1,2,4,8 and 12 weeks after discharge.
  hypnotherapy: One 90 minute session within 2 weeks of hospital discharge
- Self-Quit Group: patients were given brief counseling during hospitalization and were not be contacted until 26 weeks after hospitalization.
Arm/Group | Hypnotherapy | Nicotine Replacement Therapy | Hypnotherapy and Nicotine Replacement | Self-Quit Group
Number analyzed (Participants) | 41 | 39 | 38 | 37
Participants | 18 | 11 | 18 | 0
Statistical Analysis 1: Comparison: Hypnotherapy vs Nicotine Replacement Therapy; Test type: Superiority or Other; Adjusted for gender, marital status, diagnosis at enrollment; Risk Ratio (RR) = 2.0, 95% CI 2-sided [0.8 to 6.2]
Statistical Analysis 2: Comparison: Nicotine Replacement Therapy vs Hypnotherapy and Nicotine Replacement; Test type: Superiority or Other; Risk Ratio (RR) = 2.3, 95% CI 2-sided [1.2 to 10]

3. Secondary Outcome: Smoking Abstinence Rate at 12 and 26 Weeks
Description: Abstinence rates were calculated for patients hospitalized with a cardiac or a pulmonary diagnosis.
Time Frame: 12 weeks and 26 weeks after hospital discharge
Population: Abstinence comparing the 2 admitting diagnoses was similar within each arm, thus analysis for admitting diagnosis was done combining the 4 arms.
Measure: Number; unit: percentage of smoking abstinence rate
Groups:
- Smoking Abstinence Rates at 12 and 26 Weeks: Smoking status at follow-up time at 12 and 26 weeks by diagnosis status (cardiac vs. pulmonary)
Arm/Group | Smoking Abstinence Rates at 12 and 26 Weeks
Number analyzed (Participants) | 155
percentage of smoking abstinence rate
  % Quit rate for cardiac diagnosis at 12 weeks | 52.1
  % Quit rate for pulmonary diagnosis at 12 weeks | 20
  % Quit rate for cardiac diagnosis at 26 weeks | 34
  % quit rate for pulmonary diagnosis at 26 weeks | 20
Statistical Analysis 1: Comparison: Smoking Abstinence Rates at 12 and 26 Weeks; Comparison of smoking status at 12 weeks after hospitalization for a cardiac or pulmonary diagnosis; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Smoking Abstinence Rates at 12 and 26 Weeks; Comparison of smoking stars at 26 weeks after hospitalization for a cardiac or a pulmonary illness; Test type: Superiority or Other; p = 0.07, ANOVA

ADVERSE EVENTS:
Time Frame: 12 and 26 weeks after hospital discharge
Groups:
- Hypnotherapy: patients receiving a free intensive session of hypnotherapy within 2 weeks of hospitalization
- Nicotine Replacement Therapy: Patients receiving a free months supply of nicotine
- Hypnotherapy and Nicotine Replacement: Patients receiving hypnotherapy and nicotine supply
- Self-Quit Group: patient who decided to quit on their own
Arm/Group | Hypnotherapy | Nicotine Replacement Therapy | Hypnotherapy and Nicotine Replacement | Self-Quit Group
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/39 | 0/38 | 0/37
Other Adverse Events (participants affected / at risk) | 0/41 | 0/39 | 0/38 | 0/37

LIMITATIONS AND CAVEATS:
Comparing two vastly different modalities such as hypnosis and NRT represented a randomizing challenge, as participants and researchers could not be blinded to interventions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes